CLINICAL TRIAL: NCT03192228
Title: Evaluation of a Multidisciplinary Program of Therapeutic Education in Type 2 Diabetes Mellitus Diabetes in Order to Fix Individualized Objectives
Brief Title: Impact of a Multidisciplinary Therapeutic Education Program Being Set up for Patients With Type 2 Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier Pitie-Salpetriere (Other)
Responsible Party: Principal Investigator, Joe Elie Salem, MD, PhD, Groupe Hospitalier Pitie-Salpetriere
Other Study IDs: CIC1421-10-15
Record Dates: First submitted 2017-06-16; First posted 2017-06-20 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Diabetes Mellitus, Type 2; Patient Education as Topic
Keywords: Diabetes Mellitus, Type 2 +; Patient Education
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Treatment adequacy score — Evaluation of the program rate of success rate by a score evaluating the different criteria that the patient was supposed to modify following the therapeutic education program: practice of a physical activity, reduction of the amount of fat in Diet, practice of self-monitoring blood sugar as a motivational tool and decreased distress related to diabetes

SUMMARY:
Therapeutic education programs allows in diabetic patients to promote self-care and better perception of the disease The multidisciplinary program of therapeutic education regroups in one day: individual interview, nutritional workshop, self-monitoring blood glucose workshop, physical activity and glycemic objectives workshop.

At the end of the program, individual and personalized goals are given to the patient.

This study aims to evaluate this program success rates and the psychological, anamnesis, and sociological factors linked to success.

ELIGIBILITY:
Inclusion Criteria:

* All Type 2 diabetic patients who participate in the multidisciplinary program
* Signature information form and consent by the patient

Exclusion Criteria:

* None

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This initial education program is intended for patients with type 2 diabetes:
  * who have recently been diagnosed with type 2 diabetes
  * or who have an HbA1c greater than 7% and unability to lower their blood glucose levels despite an optimal management by general practitioner but do not yet require insulin treatment
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2012-05 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Success rate of the therapeutic education program | one month
  The rate of success of the program defined by a 50% improvement in the treatment adequacy score evaluated at 1 month

SECONDARY OUTCOMES:
Long term success rate of the therapeutic education program | 6 month
  The rate of success of the program defined by a 50% improvement in the treatment adequacy score evaluated at 6 month

IPD SHARING:
Plan to Share IPD: No